CLINICAL TRIAL: NCT06698588
Title: Examining Symptom-Specific Effects of Omega-3 Fatty Acids in Children with ADHD / ASD Symptoms and Sleep Problems: a Network Approach.
Brief Title: Symptom-specific Effects of Omega-3 Across Neurodevelopmental Symptoms
Acronym: SEASONS
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Swansea University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: Young 001
Record Dates: First submitted 2024-11-13; First posted 2024-11-21 (Actual); Last update posted 2024-11-21 (Actual); Status verified 2024-10

CONDITIONS: Sleep; Autism or Autistic Traits; ADHD or ADHD Traits
Keywords: Randomised Controlled Trial
MeSH Terms: conditions — Autistic Disorder; Attention Deficit Disorder with Hyperactivity

STUDY DESIGN:
Intervention Model Description: Whilst we are conducting an RCT we are planning on taking a modern approach to data-analysis - time-varying network analysis. This approach moves beyond the traditional medical model and its diagnostic categories where the assumption is that symptoms stem from a common underlying cause, and treating that cause (via medication or therapy) should alleviate the symptoms. This approach has been largely unsuccessful.
  In contrast, network analysis views mental health disorders as complex, interrelated systems of symptoms and does not lend itself to calculating composite of global scores (see project description for further information.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Active intervention (Experimental): Supplement
  Interventions: Dietary Supplement: Omega 3 Fish Oil supplements
- Placebo intervention (Experimental): Supplement
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Omega 3 Fish Oil supplements — Wileys Easy Swallow Mini Softgel capsules, dose 3 caps/day, providing 945mg/day long-chain omega-3 (540mg EPA, 405mg DHA).
  Arms: Active intervention
Dietary Supplement: Placebo — Placebo: high-oleic sunflower oil (which broadly matches the overall fatty acid composition of typical UK diet), matched with active treatment for appearance and taste.
  Arms: Placebo intervention

SUMMARY:
Our study aims to determine whether omega-3 fatty acid supplementation can improve sleep, mood, and behavior in children with sleep problems and symptoms of Autism Spectrum Disorder (ASD), Attention-Deficit/Hyperactivity Disorder (ADHD), or both. By using a transdiagnostic approach-focusing on specific symptoms rather than diagnostic labels-we aim to identify which children may benefit most from omega-3 supplementation, thereby enhancing inclusivity. Many previous studies have excluded children with both ASD and ADHD, or those without a formal diagnosis.

DETAILED DESCRIPTION:
ASD and ADHD are highly diverse neurodevelopmental conditions with significant co-occurrence-some estimates suggest rates as high as 78% (Leitner, 2014). However, research often excludes neurodiverse children with co-occurring conditions or subclinical symptoms, making many study populations unrepresentative of real-world scenarios. Currently, there are no fully safe and effective treatments for ASD or ADHD symptoms (Groom & Cortese, 2022; Oono et al., 2013; Williams et al., 2010), which leads many parents to explore complementary treatments, such as omega-3 supplements, among the most popular options (Green et al., 2006; Sinha & Efron, 2005). Omega-3s, essential for brain development and function, are often deficient in UK children, particularly those with behavioral or learning difficulties (Montgomery et al., 2014).

Some clinical trials suggest that omega-3 supplementation, specifically EPA (eicosapentaenoic acid) and DHA (docosahexaenoic acid), can improve symptoms such as sleep disturbances, hyperactivity-impulsivity, and inattention in children with ADHD and/or ASD-like difficulties (Bent et al., 2014; Richardson & Montgomery, 2005). However, findings across studies have been inconsistent, with systematic reviews and meta-analyses yielding varied conclusions (Abdullah et al., 2019; Bloch & Qawasmi, 2011; Gillies et al., 2012). These discrepancies likely arise from variations in study populations, treatments, outcome measures, and trial designs.

A key limitation is the traditional approach of treating ASD and ADHD as distinct diagnostic categories, adhering to the "latent variable" model in psychiatry, which assumes that symptoms reflect an underlying disorder. This approach has two major flaws: (a) it encourages studying groups presumed homogeneous based on diagnosis, ignoring within-group variability and symptom overlap across disorders, and (b) it directs treatment toward presumed underlying diseases rather than focusing on specific symptoms and their interactions. This "one-size-fits-all" model may contribute to the inconsistent findings in omega-3 research for neurodevelopmental conditions.

In contrast, network science offers a more dynamic approach, viewing disorders as networks of interacting symptoms rather than symptoms being caused by a single underlying disorder. This approach enables visualization of symptom networks, including complex connections that explain symptom overlap. For instance, "bridge" symptoms link different disorder domains, while "central" symptoms, which are highly connected, drive other symptoms and may be ideal treatment targets. Monitoring symptom networks during treatment can help identify individuals more likely to benefit based on unique symptom profiles (Bringmann et al., 2022; Bekhuis et al., 2018).

To date, the network approach has not been used to explore how omega-3 supplementation affects ASD and ADHD symptoms. Our study aims to apply this method to: (a) better understand the shared features of ADHD and ASD by identifying "bridge symptoms" and examining whether omega-3 supplementation influences these symptoms; (b) identify phenotypes that cross diagnostic boundaries and might benefit from omega-3 supplementation; and (c) promote a more inclusive approach to treating ADHD/ASD symptoms by focusing on symptom profiles rather than diagnostic labels.

We hypothesize that sleep disturbances and emotional dysregulation will act as "bridge nodes" that connect ADHD and ASD, given their presence across multiple disorders. Based on prior studies (Montgomery et al., 2014; Richardson, 2006; Richardson & Montgomery, 2005), we also propose that omega-3 supplementation will directly improve a cluster of symptoms related to sleep, emotional regulation, and hyperactivity-impulsivity. Any additional benefits are expected to be indirect, resulting from improvements in these key symptoms.

ELIGIBILITY:
Inclusion Criteria:

Autism Spectrum Quotient 10 score >5 OR Conners 3 Handscored Short Parent Form T score > 64 for either the inattention OR hyperactivity subscales OR Children Sleep Habits Questionnaire SF score >30 Able to swallow capsules

Exclusion Criteria:

Any major psychiatric condition likely to require hospitalization (e.g., Psychotic Disorders; Eating Disorders), but NB: for representativeness of typical children with ADHD/ASD, diagnosed mood/anxiety/sleep or other neurodevelopmental disorders will not be exclusion criteria; Severe learning difficulties (e.g., Down syndrome) Any serious medical condition; (d) allergy to any ingredients of the intervention or related substances

Ages: 5 Years to 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 200 (Estimated)
Dates: Start 2024-11-07 (Actual); Primary Completion 2025-06-01 (Estimated); Study Completion 2025-12-01 (Estimated)

PRIMARY OUTCOMES:
Changes in the network structure of symptoms before and after intervention. | Baseline and after 12-weeks
  This involves identifying shifts in symptom interconnectivity, which can indicate improvements in symptom clustering (e.g., a reduction in connections around "bridge" symptoms like emotional dysregulation or sleep disturbances). All questionnaires mentioned in secondary outcomes are used in the network.

SECONDARY OUTCOMES:
Autism Spectrum Quotient 10 | Baseline and after 12-weeks
  Linear mixed model - For comparison with other trials that investigated Omega 3 on ASD symptoms
Conners 3 Handscored Short Parent Forms | Baseline and after 12-weeks
  Linear mixed model - For comparison with other trials that investigated Omega 3 on ADHD symptoms including Inattention; Hyperactivity; Executive Functioning; Defiance/Aggression; Peer relations
Childrens Sleep Habits Questionnaire - SF | Baseline and after 12-weeks
  Linear mixed model - For comparison with other trials that investigated Omega 3 on sleep
Strengths and Difficulties Questionnaire | Baseline and after 12-weeks
  Linear mixed model - For comparison with other trials that investigated Omega 3 on emotional problems including Emotional symptoms; Conduct problems; Hyperactivity/inattention; Peer relationship problems; Prosocial behavior
Griffith Empathy Scale | Baseline and after 12-weeks
  Linear mixed model - For comparison with other trials that investigated Omega 3 on cognitive empathy and affective empathy
Child Mania Rating Scale Parent version | Baseline and after 12-weeks
  Linear mixed model - For comparison with other trials that investigated Omega 3 on mania
Moods and feelings Questionnaire - SF | Baseline and after 12-weeks
  Linear mixed model - For comparison with other trials that investigated Omega 3 on mood

OTHER OUTCOMES:
Arrow flanker | Baseline and after 12-weeks
  Online tests
Stop signal task | Baseline and after 12-weeks
  Online tests

CONTACTS AND LOCATIONS:
Locations (1):
- FHMLS, Swansea, United Kingdom

IPD SHARING:
Plan to Share IPD: Undecided